CLINICAL TRIAL: NCT05724888
Title: Physical Activity and Cardiovascular Disease (CVD) in Adolescents With Type 2 Diabetes: A Pilot Randomized Trial
Brief Title: Physical Activity and CVD in Adolescents With Type 2 Diabetes
Acronym: CVD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Manitoba (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other); Children's Hospital Research Institute of Manitoba (CHRIM) (Unknown)
Responsible Party: Principal Investigator, Jon McGavock, Principal Investigator, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HS25697(B2022:099)
Record Dates: First submitted 2022-12-22; First posted 2023-02-13 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Cardiovascular Diseases; Type2diabetes
Keywords: resilience; peer mentorship
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants will be from 2 different locations. 1) Winnipeg, MB, Canada 2) St. Theresa Point First Nations, MB, Canada. 20 participants will be recruited from each location and then at each location participants will be randomized in a 1:1 fashion to one of two arms for 12 weeks: (A) A behavioural lifestyle intervention that supports increased PA or (B) a control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention_Winnipeg (Experimental): The intervention arm will take place in a 12 week intervention (3 sessions per week) which will use a peer mentoring network based on the circle of courage to encourage adolescents with T2D to achieve the WHO recommended target of 300 minutes of moderate to vigorous PA weekly.
  Interventions: Behavioral: Peer mentorship and physical activity
- Control_Winnipeg (No Intervention): The control group will receive standard recommendations for increasing daily PA from the Canadian Society of Exercise Physiology and the American Heart Association.
- Intervention_STP (Experimental): The intervention arm will take place in a 12 week intervention (3 sessions per week) which will use a peer mentoring network based on the circle of courage to encourage adolescents with T2D to achieve the WHO recommended target of 300 minutes of moderate to vigorous PA weekly.
  Interventions: Behavioral: Peer mentorship and physical activity
- Control_STP (No Intervention): The control group will receive standard recommendations for increasing daily PA from the Canadian Society of Exercise Physiology and the American Heart Association.

INTERVENTIONS:
Behavioral: Peer mentorship and physical activity — Participants will be asked to participate for 12 weeks, attending 3 sessions per week (if in the intervention arm). Session 1 will be a group session that will be about 90 minutes, session 2 will be an individual session with a peer mentor for 20-30 minutes, and session 3 will be a virtual check in with the peer mentor about 15 minutes. The intervention will focus on increasing physical activity through the circle of courage.
  Arms: Intervention_STP; Intervention_Winnipeg

SUMMARY:
The main research questions for this study are: (1) Is delivering a resiliency-informed behavioural intervention designed to increase physical activity (PA) feasible for adolescents living with Type 2 Diabetes (T2D)? and (2) What is the expected change in proposed cardiovascular outcomes after 12 weeks in both study arms? Qualitative and quantitative methods embedded in this pilot randomized trial will answer these questions and determine the feasibility of a larger randomized controlled trial.

DETAILED DESCRIPTION:
Forty adolescents with T2D, 14-17 years old with a body mass index (BMI) Z score > 1.6 and do not engage in regular PA (< 300 mins of moderate to vigorous PA weekly) will be recruited from the iCARE cohort study and the pediatric T2D clinic in Winnipeg. A research assistant will recruit participants from the pediatric endocrinology clinic (DER-CA), and the Manitoba-based iCARE cohort who have previously given consent to be approached for other studies. Participants will be screened by a pediatric endocrinologist to ensure they meet inclusion criteria prior to being approached to participate. Adolescents that are eligible with be consented by the research assistant, then randomized to study arms using a computer-generated program developed by a statistician not affiliated with the study.

The control arm will receive standard recommendations for increasing daily PA from the Canadian Society of Exercise Physiology and the American Heart Association. The intervention arm will take place in a 12 week intervention (3 sessions per week) which will use a peer mentoring network based on the circle of courage to encourage adolescents with T2D to achieve the WHO recommended target of 300 minutes of moderate to vigorous PA weekly.

Session #1: Will be a group-based activity session, where adolescents will meet in person or join virtually to complete 20-30 minutes of reflecting on the past week and goal setting for upcoming week with an additional 30 to 40 minutes of PA led by a kinesiologist and peer mentor. Session #2: Will be a 15-minute wellness check, to determine emotional, mental, physical and social well-being with a peer mentor. The adolescent with T2D will also reflect on the goals set for the week and complete a structured 30-minute activity session. Session #3: Will be a 30-minute session by the adolescent on a weekend day. Prior to the session the adolescent will receive a text or social media prompts from the kinesiologist or peer mentor.

All weekly sessions throughout the 12-week intervention will incorporate the four core tenets of the Circle of CourageTM and three tenets of Self Determination Theory. During Phase 1 (Weeks 1-3) of the intervention, the focus will be on creating a sense of Belonging and relatedness. Group sessions will focus on sharing past experiences with behaviour change, unique challenges of living with T2D and shared interests or passions that will connect adolescents to each other and the intervention. During Phase 2 (Weeks 4-6), the intervention will focus on the concepts of Mastery and competence. The kinesiologist and peer mentor will encourage adolescents to focus on strengths in their lives. Reflecting on the previous four weeks and their adolescence, what behaviours or support have helped them adopt a more active lifestyle. Adolescents will also be taught land/nature-based activities by local experts as a pilot to determine appropriateness and feasibility for a larger trial. The investigators have previously demonstrated that land/outdoor-based activities are associated with significantly higher PA among adolescents. During Phase 3 (Weeks 7-9), the kinesiologist and peer mentor will foster a sense of Independence and autonomy. Adolescents will set goals, begin the process of journaling their experiences and factors that influence their motivation and actions towards adopting a more active lifestyle. During Phase 4 (weeks 10-12) the group will incorporate Generosity into their activity goals. The group will identify opportunities to be active in their communities while also giving back in some way (volunteering for Meals on Wheels, park maintenance, organize activities for children).

ELIGIBILITY:
Inclusion Criteria:

* 14-17 years old
* BMI z score >1.6
* diagnosed with type 2 diabetes

Exclusion Criteria:

* engage in >300 minutes of moderate-vigorous physical activity per week
* have diabetes because of surgery or medications for another condition
* use chronic high dose steroids or immunosuppressive therapy
* they have cancer
* the have evidence of drug or alcohol abuse
* if youth and/or parent/guardian are unable or unwilling to give consent

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-12-20 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
Enrollment rates | 12 weeks
  Defined as the number of adolescents who consent to participate and are randomized to one of the two study arms.
Adherence to the intervention arms | 12 weeks
  Defined as the percentage of prescribed sessions that adolescents/families attended during the trial.
Retention for follow-up measurements | 24 weeks
  Defined as the number of adolescents who complete follow-up measurements at randomization.

SECONDARY OUTCOMES:
Physical activity | week 1, week 12, week 24 (3 weeks total)
  Daily moderate to vigorous PA, will be assessed using 7-day waist mounted accelerometery (Actigraph). Adolescents will be asked to wear the accelerometers for 12 hours/day, seven days/week.
Readiness for behavior change | week 1, week 12, week 24 (measures will be taken at 3 different time points)
  This will be assessed using the PACE readiness questionnaire, which assesses readiness for, physical activity goals and screen time.
BREQ2 (Behavioral Regulation in Exercise Questionnaire-2) change | week 1, week 12, week 24 (measures will be taken at 3 different time points)
  the BREQ2 (Behavioral Regulation in Exercise Questionnaire-2), which is a measure of the level of motivation to engage in exercise from a self-determination perspective.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manitoba / Children's Hospital Research Institute of Manitoba (CHRIM), Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No